CLINICAL TRIAL: NCT06539572
Title: Perception of Appearance and Social Acceptance Between Cleft and Non-Cleft Children in Early Adolescence: Questionnaire Analysis Based on 3dMD Images
Brief Title: Perception of Appearance and Social Acceptance Between Cleft and Non-Cleft Children in Early Adolescence
Acronym: Cleft social
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pang-Yun Chou, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202200698B0
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cleft Lip and Palate; Social Isolation
Keywords: Cleft lip and palate; three-dimensional image technique; adolescent peers; aesthetic evaluation; psychosocial impact
MeSH Terms: conditions — Cleft Lip; Social Isolation | interventions — Alveolar Bone Grafting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cleft lip and palate: Cleft lip and palate patients, undergone surgical treatment and received regular follow-ups in the Chang Gung Craniofacial Center; aged 10-12; after alveolar bone grafting surgery
  Interventions: Procedure: Cleft lip repair; palatoplasty; alveolar bone grafting
- Non-cleft: Non cleft cohort as control group; recruited from various elementary schools in the Guishan district of Taoyuan City, Taiwan; aged 10-12; without craniofacial anomalies.

INTERVENTIONS:
Procedure: Cleft lip repair; palatoplasty; alveolar bone grafting — cleft surgical treatment based on Chang Gung Craniofacial Center Protocol for cleft treatment
  Groups: Cleft lip and palate

SUMMARY:
Background: Using three-dimensional (3D) surface imaging, this study aims to understand the differences in perception between schoolchildren with and without cleft lip and palate (CLP), as well as to explore peer awareness and acceptance of children with craniofacial abnormalities post-surgery.

Methods: This cross-sectional study utilized three-dimensional surface images of early adolescent patients with CLP post-repair and without CLP for examination by schoolchildren (with CLP and without). Both groups assessed the images and responded to a questionnaire eliciting perceptions of facial appearance and social acceptance of children with craniofacial abnormalities, rating each question on a Likert scale of one to five. The results were presented using bar graphs, and the Item Response Theory-Graded Response Model was employed to estimate the latent ability (θ) of each participant. The reliability of the questionnaire was assessed with Cronbach's alpha test.

ELIGIBILITY:
Inclusion Criteria:

* Cleft patient received cleft surgical treatment including lip repair, palatoplasty, and alveolar bone grafting in our Craniofacial Center, based on our cleft surgical protocol

Exclusion Criteria:

* Unable to complete the questionnaire on their own for any reason were excluded to avoid bias in responses caused by the presence of a secondary observer

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: <Acquisition of 3D Image>
  * Cleft: Images of subjects with and without craniofacial anomalies were extracted from the database at the Chang Gung Craniofacial Research Center; taken before and after alveolar bone graft surgery at a six-month interval, from 2017 to 2020; aged about 9.
  * Noncleft: healthy pediatric individuals from six to 12 years of age. Randomly selected from the database, aged 9-12
  <Participants for questionnaires>
  * CLP patients and non-cleft children aged 10-12 were randomly recruited
  * Patients with CLP were sourced from individuals who had undergone surgical treatment and received regular follow-ups in our Craniofacial Center; the non-cleft cases were recruited from various elementary schools in the Guishan district of Taoyuan City, Taiwan.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Facial appearance | 6 months after alveolar bone grafting
  based on 3dMD image

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No